CLINICAL TRIAL: NCT06817291
Title: Laparoscopic Endobiliary Stent and Postopertive ERCP Compared to Intraoperative ERCP for the Treatment of Common Bile Duct Stones: A Swedish Registry Bases Study
Brief Title: Laparoscopic Endobiliary Stent and Postoperative ERCP Compared to Intraoperative ERCP
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Camilla Runfors, MD, PhD, Karolinska Institutet
Other Study IDs: 2023-05310-01
Record Dates: First submitted 2025-01-24; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Common Bile Duct Stones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Laparoscopic endobiliary stent and postponed ERCP: Intraoperatively found common bile duct stones treated with laparoscopic endobiliaty stent and postoperative ERCP
  Interventions: Procedure: Laparoscopic endobiliary stent
- Intraoperativ ERCP: Intraoperatively found common bile duct stones treated with intraoperative ERCP

INTERVENTIONS:
Procedure: Laparoscopic endobiliary stent — During laparoscopic gallblader surgery, a quidewire is inserted in the cystic duct, via the common bile duct and advanced into the duodenum. The plastic stent is threaded over the wire and pushed in position, with a catheter. When the stent is crossing the papilla, the wire is first removed, and then the catheter. The procedure is done under x-ray guidance.
  Groups: Laparoscopic endobiliary stent and postponed ERCP

SUMMARY:
Laparoscopic endobiliary stent and postponed endoscopic retrograde cholangiopancreatography, ERCP, compared to intraoperative ERCP for the treatment of common bile duct stones, CBDS, a retrospective registry based cohort study.

Data will be collected from GallRiks, the Swedish national registry for cholecystectomies and ERCP. Patients in the registry identified with found of CBDS at intraoperative cholangiography, IOC, and there after treated with ERCP during 2010-01-01 to 2023-12-31 are the study population.

Research question: In patients with intraoperatively diagnosed CBDS - is there a difference in complications between laparoparoscopic endobiliary stent with postoperative ERCP, and intraoperative ERCP? Primary outcome: Complications within 30 days after cholecystectomy and the following ERCP.

Secondary outcomes: 30 day mortality, procedure time for cholecystectomy, procedure time for ERCP, difficult cannulation, stone clearance at ERCP, cumulative hospital stay, readmission within 30 days after cholecystectomy/ERCP

DETAILED DESCRIPTION:
In Sweden, the common bile duct is routinely examined during cholecystectomy, by using radiography with a contrast agent, IOC. Arguments for IOC are to clarify the anatomy, to detect possible bile duct injury, and to reveal stones in the CBD. Today many cholecystectomies in Sweden are performed in units with no or limited access to ERCP. In these cases, intraoperative ERCP is not always a viable option. Placing an endobiliary stent is an alternative when CBD stones are found intraoperatively by cholangiography. A guidewire can be inserted via the cholangiography-catheter (already placed in the duodenum after IOC), to the CBD, and further on into the duodenum. A plastic stent is then inserted over the wire. The stent is positioned to extend from the CDB into the duodenum. The endobiliary stent prevents bile obstruction from stones in the CBD. Subsequent ERCP, to remove stent and stones, can be postponed to a couple of weeks after the cholecystectomy. Endobiliary stents have been used to a smaller extent in Sweden since the 90s. Observational studies have described facilitation of cannulation during postoperative ERCP if an endobiliary stent has been placed.

Earlier studies publiched includes less than a hundred patients.

By using Swedish national registry data from GallRiks it will be possible to inlcude more patients then previsus studies with endobiliary stent, and also have a comparison group.

The study will compare morbidity with the treatment strategy endobiliary stent and postoperative ERCP to intraoperative ERCP. Intraoperative ERCP is gold standard in Sweden for management of CBDS found intraoperatively. Morbidity includes complications within 30 days from cholecystectomy and 30 days from ERCP.

There is a need to manage CBD stones detected during IOC in a safe and effective manner, even when intraoperative ERCP cannot be performed. Endobiliary stent is used in clinical practice today, and could be used to a larger extent, and become a valuable contribution in CBDS treatment, if the method would gain stronger scientific support.

ELIGIBILITY:
Inclusion Criteria:

Laparoscopic choleystectomy with intraoperative found of common bile duct stones by intraoperative cholangiography.

Common bile duct treated with laparoscopic endobiliary stent and postponed ERCP or intraoperative ERCP

Exclusion Criteria:

Other types of treatment for common bile duct stones Conversion to or open cholecystectomy

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will be identified in the GallRiks registry with found of CBDS at intraoperative cholangiography, IOC, and thereafter treated with ERCP during 2010-01-01 to 2023-12-31.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Complication after cholecystectomy and the following ERCP | 30 days after each procedure
  Number of participants with treatment-related adverse events such as pancreatitis, cholangitis, bleeding, infection, gall leakage

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Sciences, Danderyd Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No